CLINICAL TRIAL: NCT00043745
Title: Bone Response to Soy Isoflavones in Women
Acronym: SIRBL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01AR046922 (NIH); R01AR046922 (NIH); NIAMS-073
Record Dates: First submitted 2002-08-13; First posted 2002-08-14 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Osteopenia; Osteoporosis
Keywords: soy; isoflavones; alternative hormone therapy; bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive moderate dose soy isoflavone (80 mg/day) tablets, extracted from soy protein
  Interventions: Dietary Supplement: Soy isoflavones
- 2 (Experimental): Participants will receive high dose soy isoflavone (120 mg/day) tablets, extracted from soy protein
  Interventions: Dietary Supplement: Soy isoflavones
- 3 (Placebo Comparator): Participants will receive soy extract devoid of isoflavones to serve as placebo
  Interventions: Dietary Supplement: Extract tablets

INTERVENTIONS:
Dietary Supplement: Soy isoflavones — Soy isoflavones extracted from soy protein, compressed into tablets; three tablets taken daily
  Arms: 1; 2
Dietary Supplement: Extract tablets — Extract from soy protein, but devoid of isoflavones; three tablets taken once daily
  Arms: 3

SUMMARY:
This study will provide valuable data on whether soy isoflavones impact bone loss in postmenopausal women. The study will help clarify potential mechanisms and contribute to our understanding of isoflavones as an alternative to traditional hormone therapy.

DETAILED DESCRIPTION:
Soy protein, rich in isoflavones (estrogen-like compounds), has been shown to prevent bone loss in ovariectomized rats. Short-term preliminary study results in perimenopausal women suggest a bone-sparing effect. Great interest in isoflavones as an alternative to hormone replacement therapy has emerged, yet the long-term efficacy of isoflavones on bone in humans is unknown. Our objective is to determine the three-year efficacy of isoflavone-rich soy extract in attenuating bone loss in postmenopausal women. The central hypothesis is that soy isoflavones will attenuate bone loss in these women by maintaining bone formation, which is modulated by growth factors and isoflavone metabolism. The rationale for this research is that current hormone therapy is fraught with adverse side effects, resulting in non-compliance. This randomized, double-blind, placebo-controlled clinical trial will examine the effects of two doses (80 or 120 mg daily) of isoflavone-rich soy extract on bone in non-osteoporotic postmenopausal women (N=234). The specific aims of this study are: 1) to determine the bone-preserving effects of isoflavones on lumbar spine bone mineral density (BMD); 2) to relate treatment-induced changes in BMD to changes in biochemical markers of bone turnover; 3) to identify potential mechanisms by which isoflavones prevent or modulate bone loss by measuring endogenous estrogens, sex hormone-binding globulin, insulin-like growth factor-I (IGF-I), urinary minerals, serum 25(OH)vitamin D, plasma isoflavones and their metabolites, and customary intake of isoflavone-containing soy; and, 4) to ascertain the safety of isoflavone-rich soy extract. Postmenopausal women will be recruited at two sites (117 at Iowa, 117 at California). Random effects repeated measures analyses will be used to characterize change in BMD as the primary outcome, estimate treatment-induced effects, and depict change in markers of bone turnover in relation to BMD change. We will use intent-to-treat for the primary test, but also account for potential modulators (reproductive hormones, IGF-I, plasma isoflavones) that affect bone, as indicated in specific aim 3.

ELIGIBILITY:
Inclusion Criteria:

* Early postmenopausal (i.e., no menses during past 12 months) women, with an upper limit of 10 years since their last cycle
* Natural menopause (i.e., no hysterectomies or oophorectomies)
* Body mass index (BMI) > 20 and < 30

Exclusion Criteria:

* Current or previous (within 12 months) use of hormone replacement therapy, hormonal contraceptives, estrogens, or progestogens
* Current use of pharmacologic agents, such as selective estrogen-receptor modulators (SERMs) (e.g., raloxifene or tamoxifen) or anti-resorptive agents (e.g., alendronate or calcitonin), herbal therapies that may have estrogenic effects (e.g., herbimycin, tryphostins), or cigarettes
* Strict vegans (but will include lacto-ovo-, lacto-, and ovo-vegetarians)
* Metabolic bone disease, renal disease, history of urolithiasis, cancer, cardiovascular disease, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease, or other chronic diseases
* First-degree relative with breast cancer
* Lumbar spine BMD >= -1.5 standard deviations (SD) below mean (high-risk for osteoporosis) and BMD >= +1.0 SD above mean

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2003-03; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Lumbar spine bone mineral density | Year 3

SECONDARY OUTCOMES:
Proximal femur bone mineral density | Year 3

CONTACTS AND LOCATIONS:
Overall Officials: D. Lee Alekel, PhD, Principal Investigator — Iowa State University
Locations (2):
- United States (2):
  - USDA/ARS/WHNRC University of California-Davis, Davis, California
  - Iowa State University, Ames, Iowa

REFERENCES:
- [Derived] Alekel DL, Genschel U, Koehler KJ, Hofmann H, Van Loan MD, Beer BS, Hanson LN, Peterson CT, Kurzer MS. Soy Isoflavones for Reducing Bone Loss Study: effects of a 3-year trial on hormones, adverse events, and endometrial thickness in postmenopausal women. Menopause. 2015 Feb;22(2):185-97. doi: 10.1097/GME.0000000000000280. PMID 25003624
- [Derived] Matvienko OA, Alekel DL, Genschel U, Ritland L, Van Loan MD, Koehler KJ. Appetitive hormones, but not isoflavone tablets, influence overall and central adiposity in healthy postmenopausal women. Menopause. 2010 May-Jun;17(3):594-601. doi: 10.1097/gme.0b013e3181c92134. PMID 20142790
- [Derived] Alekel DL, Van Loan MD, Koehler KJ, Hanson LN, Stewart JW, Hanson KB, Kurzer MS, Peterson CT. The soy isoflavones for reducing bone loss (SIRBL) study: a 3-y randomized controlled trial in postmenopausal women. Am J Clin Nutr. 2010 Jan;91(1):218-30. doi: 10.3945/ajcn.2009.28306. Epub 2009 Nov 11. PMID 19906801